CLINICAL TRIAL: NCT03499093
Title: Development and Validation of the French Version of the Orofacial Esthetic Scale: OES-F
Brief Title: French Version of the Orofacial Esthetic Scale
Status: Completed | Type: Observational
Sponsor: Hôpital Rothschild (Other)
Responsible Party: Principal Investigator, Dr Braud Adeline, Lecturer in odontology-hospital practitioner, Hôpital Rothschild
Other Study IDs: 2016/303 (2)
Record Dates: First submitted 2018-03-28; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Esthetics, Dental
Keywords: esthetics; orofacial esthetic scale
MeSH Terms: interventions — Moire Topography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Prosthetic patient with esthetic expectations: Prosthetic patients with esthetic expectations (PP-E, n=35), Patients seeking for restoration or replacement of anterior teeth, or expressing any esthetic expectation
  Interventions: Other: OES
- Prosthetic patients without esthetic expectations: Prosthetic patients without esthetic expectations (PP-NE, n=35) Patients pending restoration or replacement of posterior teeth (premolars and molars), expressing only functional expectation
  Interventions: Other: OES
- Dental patient with esthetic concern: Dental patient with esthetic concern(C-E, n=35) Patient consulting for follow up, having crowns or removable denture replacing anterior teeth
  Interventions: Other: OES
- Dental patient without any esthetic concern: Dental patient without any esthetic concern (C-NE, n=35) Patient consulting for follow up, having no crown or removable denture replacing anterior teeth.
  Interventions: Other: OES

INTERVENTIONS:
Other: OES — The first seven items of OES refer to face, facial profile, mouth, teeth alignment, teeth form, teeth color and gums. They are combined into an OES summary score ranging from 0 to 70. The eight item of OES is an overall impression item and is not included in the summary score.
  Internal Consistency was determined using Cronbach's alpha and inter-item correlation for the OES scores (n=140).
  Test-Retest Reliability was assessed using Intraclass Correlation Coefficient. Patients with prosthetic needs (n=20 PP-E subjects and n=15 PP-NE subjects) completed twice the OES-F at an interval of two weeks.
  Convergent validity was assessed by comparing mean OES summary scores evaluated by participant of the esthetic group (PP-E, n=35) and by an expert group. Expert OES score were based on three photographs of each participant.
  Discriminative validity was tested by comparing the OES summary scores using a one-way ANOVA and Scheffe post hoc test.
  Other Names: Photographs

SUMMARY:
The aims of this study were to develop a French version of the Orofacial Esthetic Scale (OES-F) and to investigate its psychometric properties.

The OES is an eight-item instrument that assesses self-reported orofacial esthetics in prosthodontic patients. The first seven items refer to direct esthetic impacts and the eight is a global assessment item. For each item, an 11-point numeric scale (ranged from 0 = very dissatisfied to 10 = very satisfied) is used, and the first seven scores are combined into a summary score from 0 (worst score) to 70 (best score). The original English version of the OES was translated into French according to the guidelines. The reliability (internal consistency and test-retest reliability) and validity (convergent and discriminative validities) were tested in a sample of 140 patients. To assess test-retest reliability, 35 patients answered twice the OES-F with a temporal distance of two weeks apart.

DETAILED DESCRIPTION:
Participants From September 2016 to december 2017, 160 patients aged over 18 have been recruited at the university dental clinic of the Rothschild Hospital, Paris, among patients pending dental treatment. Inclusion criteria were : literate French speakers, willing and able to complete the survey in a single setting. Patients suffering from head and neck tumors, defects after tumor resection, radiotherapy treatment, patients suffering from dementia or cognitive impairment, and communication difficulties were excluded.

The pilot version was tested in a sample of twenty patients who were not involved in the main study. One hundred forty patients answered the final French version of the questionnaire to assess the psychometric properties of the OES-F. They were first divided into two groups according to their prosthetic needs. Participants were further allocated to two groups according to their esthetical concerns. Finally, the french version of the OES was tested with n=35 prothetic patients with esthetic expectations (PP-E), with n=35 prothetic patients without esthetic expectations (PP-NE), with n=35 subjects with esthetic concerns (C-E) and n=35 subjects without any esthetic concern (C-NE). Prosthetic patients were recruited either during the initial visit or before prosthetic treatment. Control subjects were recruited either during their initial visit or a follow-up consultation.

All subjects provided written informed consent before inclusion and had their anonymity respected throughout the course of the study. The study was approved by the Ethics Committee of research projects of the Robert Debré Hospital (n° 2016/303(2). In application of the french law of January 6, 1978 relative to information technology, the study has been declared to the national data protection agency under the number 1977961v0.

Development of the french OES version The traduction and cross-cultural adaptation was performed according to the guidelines. Briefly, the english version was first translated into french by two dental practitioners and then back translated in english by two native english speakers. Both translated versions were discussed by the research team and appropriate changes were formulated to the french version if necessary to clarify any item of the questionnaire. Clear understanding of any question and the entire french version of the questionnaire was tested with twenty participants. Minor changes concerned only formulation of general presentation of the questionnaire.

The psychometric validity of the final french version was finally tested, including reliability and validity.

ELIGIBILITY:
Inclusion Criteria:

* literate French speakers, willing and able to complete the survey

Exclusion Criteria:

* Patients suffering from head and neck tumors, defects after tumor resection, radiotherapy treatment, patients suffering from dementia or cognitive impairment, and communication difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients pending dental treatment or follow up at the university dental clinic of the Rothschild Hospital, Paris.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline orofacial esthetic scale (OES) summary score at two weeks | evaluated at date of inclusion and two weeks later
  The first seven items refer to esthetic components: face, facial profile, mouth (smile, lips, and visible teeth), teeth alignment, teeth form, teeth color and gums. These seven scores are combined into an OES summary score ranging from 0 (worst score, patient is very dissatisfied with all esthetics items) to 70 (best score, patient is very satisfied with all esthetics items).

SECONDARY OUTCOMES:
Change from baseline overall impression (eight item of OES questionnaire) at two weeks | evaluated at date of inclusion and two weeks later
  The eight item is an overall impression item and is not included in the summary score.

IPD SHARING:
Plan to Share IPD: No